# Time for a Diagnostic Paradigm Shift From STEMI/NSTEMI to OMI/NOMI (DIFOCCULT-3)

NCT06570759 June 29th, 2024

# Kimlik Bilgileri (Identification)

| Study ID# | |
|---|---|
| National ID# | |
| Has the patient been excluded ? | ○ Evet<br>○ Hayır |
| The reason for exclusion | <ul> <li>An alternative cause for troponin elevation</li> <li>Pregnancy or suspicion of pregnancy</li> <li>Reperfused by thrombolytic therapy instead of PC</li> <li>Rejection or withdrawal of consent</li> <li>Unable to retrieve pre-PCI ECGs</li> <li>Other</li> </ul> |
| If other is chosen, please explain. (Please briefly explain the reason for exclusion.) | 2 |
| Name and surname | |
| (e.g.; John Doe) | |
| Age | |
| Gender | ○ Male ○ Female |
| Boy<br>(in centimeters) | |
| Kilo<br>(in kilograms) | |
| Phone number<br>(Required for follow-up. E.g; 0532 510 97 98, 0216<br>283 38 38) | |
| Second phone number (if possible)<br>(Recommended for follow-up. E.g.; 0532 510 97 98, 0216 283 38 38) | |



# Randomizasyon (Randomization)

| Study ID# | |
|---|---|
| Conton | O Arthur Edit City Hearital |
| Center | <ul> <li>Ankara Etlik City Hospital</li> <li>Antalya City Hospital</li> <li>Bagcilar Training and Research Hospital</li> <li>Dasaksehir Pine and Sakura City Hospital</li> <li>Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital</li> <li>Erzurum Ataturk University, Faculty of Medicine</li> <li>Eskisehir Osmangazi University</li> <li>Eskisehir City Hospital</li> <li>Kartal Kosuyolu High Specialization Education and Research Hospital</li> <li>Kütahya Health Sciences University</li> <li>Marmara University, Pendik Training and Research Hospital</li> <li>Mehmet Akif Ersoy Training and Research Hospital</li> <li>Mugla Sitki Kocman University</li> <li>Necmettin Erbakan Meram Faculty of Medicine</li> <li>Sirnak State Hospital</li> <li>Tokat Gaziosmanpasa University Hospital</li> </ul> |
| | Van Training and Research Hospital Van Yuzuncu Yil Faculty of Medicine |
| Randomization date<br>(Enrollment date) | erila distrib |
| Study arm<br>(According to the team on duty) | STEMI/NSTEMI OMI/NOMI |
| Ön tanı<br>(Working diagnosis that caused to proceed to angiography o<br>diagnosis may not be necessarily with the preliminary diagno | |
| ○ ST-segment elevation MI (STEMI) ○ non-ST-segment el | evation MI (NSTEMI) Other |
| Any "very-high risk" NSTEMI feature ? | <ul> <li>☐ Hemodynamic instability or cardiogenic shock</li> <li>☐ Acute heart failure due to ischemia</li> <li>☐ Life-threatening ventricular arrhythmias or cardiac arrest</li> <li>☐ Mechanical complications (ischemic VSD, acute ischemic mitral regurgitation etc.)</li> <li>☐ Refractory or recurrent chest pain despite medical therapy</li> <li>☐ Dynamic ST-T wave changes, especially with intermittent ST-segment elevation</li> <li>☐ None of above</li> </ul> |



| Ön tanı<br>(Working diagnosis that caused to proceed to angiograph<br>diagnosis may not be necessarily with the preliminary dia | |
|---|---|
| ○ Occlusion MI (OMI) ○ Non-occlusion MI (NOMI) ○ | Other |
| Any "high risk" feature NOMI ? | <ul> <li>☐ Hemodynamic instability or cardiogenic shock</li> <li>☐ Acute heart failure due to ischemia</li> <li>☐ Life-threatening ventricular arrhythmias or cardiac arrest</li> <li>☐ Mechanical complications (ischemic VSD, acute ischemic mitral regurgitation etc.)</li> <li>☐ None of above</li> </ul> |
| Please explain<br>(Unstable angina, suspicious but nondiagnostic ECG,<br>cat lab availability, pre-planned angiography etc.) | |
| Informed consent form (Downloadable from this link, if required.) [Attachment: "Onam.pdf"] | Kijal Le |
| Upload the signed informed consent. (Only signature page is required. Keep the original.) | (Sigh in |
| Since the patient is excluded, you do not need to fill this (If you think this is an error, please check your answer for (Identification).) | form. r "Has the patient been excluded ?" on the first form |

## Özgeçmiş (Medical History)

| Study ID# | | |
|---|---|---|
| Hypertension (Average blood pressure >140/90 mmHg or use of antihypertensive medication) | ○ Evet | ○ Hayır |
| Diabetes (FPG>126 mg/dL for two times or HbA1c>%6.5 or use of antidiabetic medication) | ○ Evet | ○ Hayır |
| Dyslipidemia | ○ Evet | ○ Hayır |
| (LDL>160 mg/dL or use of antihyperlipidemic drug) | | |
| Active smoking<br>(Smoking history in the last one year) | ○ Evet | ○ Hayır |
| Chronic kidney disease<br>(GFR < 60 ml/min/1.73 m2 known or supposed to be<br>longer than 3 months) | ○ Evet | ○ Hayır |
| Prior myocardial infarct (Documented diagnosis or imaging evidence of an old [>1 month] myocardial infarct) | ○ Evet | ○ Hayır |
| Prior percutaneous coronary intervention | ○ Evet | ○ Hayır |
| (Documented history or imaging evidence of a prior coronary intervention) | | 5 |
| Prior coronary arterial by-pass grafting<br>(Documented history or imaging evidence of a prior<br>CABG) | ○ Evet | ○ Hayır |

Since the patient is excluded, you do not need to fill this form.
(If you think this is an error, please check your answer for "Has the patient been excluded?" on the first form (Identification).)



#### Randomizasyon (Randomization)

| Study ID# | |
|---|---|
| | <del></del> |
| | <ul> <li>Ankara Etlik City Hospital</li> <li>Antalya City Hospital</li> <li>Bagcilar Training and Research Hospital</li> <li>Dasaksehir Pine and Sakura City Hospital</li> <li>Dr. Siyami Ersek Thoracic and Cardiovascular Surgery Training and Research Hospital</li> <li>Erzurum Ataturk University, Faculty of Medicine</li> <li>Eskisehir City Hospital</li> <li>Kartal Kosuyolu High Specialization Education and Research Hospital</li> <li>Kütahya Health Sciences University</li> <li>Marmara University, Pendik Training and Research Hospital</li> <li>Mehmet Akif Ersoy Training and Research Hospital</li> <li>Mugla Sitki Kocman University</li> <li>Necmettin Erbakan Meram Faculty of Medicine</li> <li>Ordu State Hospital</li> <li>Sanliurfa Mehmet Akif Inan Training and Research Hospital</li> <li>Sirnak State Hospital</li> <li>Tokat Gazi Osman Pasa University Hospital</li> <li>Van Training and Research Hospital</li> <li>Van Training and Research Hospital</li> <li>Van Training and Research Hospital</li> <li>Van Yuzuncu Yil Faculty of Medicine</li> </ul> |
| Randomization date<br>(Enrollment date) | |
| Study arm<br>(According to the team on duty) | ○ STEMI/NSTEMI ○ OMI/NOMI |
| Preliminary diagnosis<br>(Working diagnosis that caused to proceed to angiography or adm | mission [whichever is the first]) |
| ST-segment Elevation Myocardial Infarction (MI) Criteria: | |
| (1) New J-point elevation according to the following cut-offs in two | o consecutive leads: |
| * In V2-V3, ≥40 males ≥ 2 mm; < 40 males ≥2.5 mm, females ≥ | :1.5 mm, |
| * in all other leads ≥1 mm | |
| * (includes V7-9 ST-segment elevation or V1-4 ST-segment depre | ssion for "posterior" MI) |
| <ul><li>(2) a peak troponin exceeding 99.percentile with a characteristic</li><li>(3) a clinical picture compatible with acute coronary syndrome.</li></ul> | increase and decrease (retrospective) |

**₹**EDCap®

projectredcap.org

| ○ ST-segment elevation MI (STEMI) ○ non-ST-segment | t elevation MI (NSTEMI) Other |
|---|---|
| Any "very-high risk" NSTEMI feature ? | <ul> <li>Hemodynamic instability or cardiogenic shock</li> <li>Acute heart failure due to ischemia</li> <li>Life-threatening ventricular arrhythmias or cardiac arrest</li> <li>Mechanical complications (ischemic VSD, acute ischemic mitral regurgitation etc.)</li> <li>Refractory or recurrent chest pain despite medical therapy</li> <li>Dynamic ST-T wave changes, especially with intermittent ST-segment elevation</li> <li>None of above</li> </ul> |
| Preliminary diagnosis<br>(Working diagnosis that caused to proceed to angiography | y or admission [whichever is the first]) |
| Kriterler: | |
| (1) ECG findings suggestive of acute coronary occlusion (c | or an OMI diagnosis by the App) |
| (2) a peak troponin exceeding 99.percentile with a characteristic | cteristic increase and decrease (retrospective) |
| (3) a clinical picture compatible with acute coronary syndi | rome. |
| OMI should be selected if proceeded to cath lab only with (retrospectively). Patients meeting only 2nd and 3rd criter | |
| Occlusion MI (OMI) Non-occlusion MI (NOMI) | Other |
| Any "high risk" feature NOMI ? | <ul> <li>Hemodynamic instability or cardiogenic shock</li> <li>Acute heart failure due to ischemia</li> <li>Life-threatening ventricular arrhythmias or cardiac arrest</li> <li>Mechanical complications (ischemic VSD, acute ischemic mitral regurgitation etc.)</li> <li>None of above</li> </ul> |
| Please explain<br>(Suspicious but nondiagnostic ECG, cat lab<br>availability, pre-planned angiography etc.) | |
| Informed consent form<br>(Downloadable from this link, if required.) | |
| [Attachment: "Onam.pdf"] | |
| Upload the signed informed consent. (Only signature page is required. Keep the original.) | |

Since the patient is excluded, you do not need to fill this form. (If you think this is an error, please check your answer for "Has the patient been excluded?" on the first form (Identification).)

#### Önceki tedavisi (Prior medication)

| Study ID# | |
|---|---|
| Aspirin<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| P2Y12 inhibitor<br>(Medications used before the admission) | <ul><li>○ None</li><li>○ Clopidogrel</li><li>○ Ticagrelor</li><li>○ Prasugrel</li></ul> |
| OAC/NOAC<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| ACEi/ARB<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| ARNI<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| SGLT2i<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| Beta-blocker<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| Calcium channel blocker<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| MRA<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| Loop diuretic<br>(Medications used before the admission) | ○ Evet ○ Hayır |
| Statin<br>(Medications used before the admission) | ○ Evet ○ Hayır |

Since the patient is excluded, you do not need to fill this form. (If you think this is an error, please check your answer for "Has the patient been excluded?" on the first form (Identification).)



# Başvuru sırasındaki klinik değişkenler (Clinical parameters on admission)

| Study ID# | |
|---|---|
| Mode of admission (Directly or by referral) | <ul><li>Directly (by themself or by ambulance)</li><li>Referred (from another institution)</li></ul> |
| NOTE: With regard to the admission to the randomizing (PCI-capable) center. | |
| Systolic blood pressure on admission (in mmHg) | |
| Heart rate on admission (in beats per minute) | |
| Killip class on admission<br>NOT: Başvurudan randomizasyonun yapıldığı hastane (ana çalış<br>kastedilmektedir. | macının çalıştığı primer PKG merkezi) |
| <ul> <li>Class 1: No evidence of heart failure</li> <li>Class 2: Pulmonary rales, S3 or increased jugular venous pre</li> <li>Class 3: Overt pulmonary edema</li> <li>Class 4: Signs of cardiogenic shock (oliguria, cyanosis, pale a mmHg)</li> </ul> | |
| Cardiopulmonary resuscitation before admission (Need for chest compressions, defibrillation or intubation before randomization) | ○ Evet ○ Hayır |
| Creatinine on admission (Just before or after randomization, in mg/dL, e.g.; 1.2) | |
| Hemoglobin on admission (Just before or after randomization, in g/dL, e.g.; 12.3) | |
| Very-high troponin level for this center is 1000 ng/L (According to the kit used by this center in ng/L [=pg/mL]. This occlusion) | level suggests a major epicardial coronary artery |
| Very-high troponin level for this center is 2400 ng/L (According to the kit used by this center in ng/L [=pg/mL]. This occlusion) | level suggests a major epicardial coronary artery |

Very-high troponin level for this center is 5000 ng/L (According to the kit used by this center in ng/L [=pg/mL]). This level suggests a major epicardial coronary artery occlusion)



| Troponin on admission (first troponin in ng/L [=pg/mL], e.g.; 12) | |
|---|---|
| NOTE: If not taken on admission, can be obtained during angiography. | |
| If present, second troponin (second troponin in the ER in ng/L [=pg/mL], e.g.; 12) | |
| Duration of pain (The duration of the last pain in minutes. If continuing, calculate the time to ECG from the onset of last constant pain.) | |
| Intermittent chest pain before MI ?<br>(Before the last infarct-related pain, did the patient<br>experience pain episodes in the previous month ?) | ○ Evet ○ Hayır |
| Upload the first ECG<br>(This may not be the diagnostic one. To upload further<br>ECGs, use additional areas below) | 3 |
| NOTE: Use image files (.jpg, .png, .tiff vb.) or pdf. | . 0 |
| or | |
| You can also use report code on PMCardio App<br>(For example, enter only 6c40a7ab for "Report<br>6c40a7ab" on PMCardio App.) | |
| {ekg1_reportno} | |
| *must provide a value. | O, |
| Time of the first ECG<br>(The date on ECG as day/month/year and hour:minute) | <u> </u> |
| Upload the second ECG<br>NOTE: Use image files (.jpg, .png, .tiff vb.) or pdf. | |
| or | |
| You can also use report code on PMCardio App (For example, enter only 6c40a7ab for "Report 6c40a7ab" on PMCardio App.) | |
| {ekg_reportno_2} | |
| *must provide a value. | |



| Upload the third ECG<br>NOTE: Use image files (.jpg, .png, .tiff vb.) or pdf. |
|---|
| or |
| You can also use report code on PMCardio App (For example, enter only 6c40a7ab for "Report 6c40a7ab" on PMCardio App.) |
| {ekg_reportno_3} |
| *must provide a value. |
| Upload the fourth ECG<br>NOTE: Use image files (.jpg, .png, .tiff vb.) or pdf. |
| or |
| You can also use report code on PMCardio App (For example, enter only 6c40a7ab for "Report 6c40a7ab" on PMCardio App.) |
| {ekg_reportno_4} |
| *must provide a value. |
| Upload the fifth ECG<br>NOTE: Use image files (.jpg, .png, .tiff vb.) or pdf. |
| or |
| You can also use report code on PMCardio App (For example, enter only 6c40a7ab for "Report 6c40a7ab" on PMCardio App.) |
| {ekg_reportno_5} |
| *must provide a value. |
| Which one of the uploaded ECGs lead to the diagnosis ? (Anter the number of the diagnostic ECG. If diagnosis was not based on ECG, enter "0") |
| Enter the time of this diagnostic ECG (Enter the time on the diagnostic ECG as day/month/year and hour:minute. This may be the same as the first ECG) |



| Was chest pain present during this diagnostic ECG (or during any of the ECGs, if none of them were diagnostic) ? | ○ Evet ○ Hayır |
|---|---|
| How many minutes is it since the last pain stopped ? | |
| (Enter the duration of pain from the cessation of the last episode to the ECG, in minutes.) | |
| Since the patient is excluded, you do not need to fill this form (If you think this is an error, please check your answer for "Ha (Identification).) | as the patient been excluded ?" on the first form |

#### EKG modülü (ECG module) Audit

| Study ID# |
|---|
| You are viewing ECGs from the patient with the record number of [record_id], who is a [age] year-old [gender]. This patient was admitted to [merkez] on [randomizasyon_tarihi]. |
| To access PMCardio App: https://difoccult.pmcardio.com |
| The first pre-PCI ECG |
| [ekg1:inline] QoH interpretation: |
| {ecgmodule_pre1qoh} |
| The second pre-PCI ECG |
| [ekg1:inline] QoH interpretation: |
| {ecgmodule_pre2qoh} |
| The third pre-PCI ECG |
| [ekg1:inline] QoH interpretation: |
| {ecgmodule_pre3qoh} |
| The fourth pre-PCI ECG |
| [ekg1:inline] QoH interpretation: |
| {ecgmodule_pre4qoh} |
| The fifth pre-PCI ECG |
| [ekg1:inline] QoH interpretation: |
| {ecgmodule_pre5qoh} |



## EKG modülü (ECG module) 1

| Study ID# | |
|---|---|
| You are viewing ECGs from the patient with the record number patient was admitted to [merkez] on [randomizasyon_tarihi]. | er of [record_id], who is a [age] year-old [gender]. This |
| To access PMCardio App: https://difoccult.pmcardio.com | |
| The first pre-PCI ECG | |
| [ekg1:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | 3 |
| The second pre-PCI ECG | 1 0 1.0 |
| [ekg2:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | ~(0) |
| The third pre-PCI ECG | |
| [ekg3:inline] | |
| Expert interpretation: | 4.65 |
| ○ OMI ○ not-OMI ○ Undefined | |
| The fourth pre-PCI ECG | |
| [ekg4:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | |
| The fifth pre-PCI ECG | |
| [ekg5:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | |
| Are there any dynamic changes suggestive of OMI in pre-PCI ECGs ? | <ul><li>Yes</li><li>No</li><li>Undefined</li></ul> |
| (Dynamic ST-T changes, Q wave development) | Officerified |
| The first post-PCI ECG | |
| [postpci_ekg:inline] | |



| Post-PCI 24h ECG | |
|---|---|
| [postekg24:inline] | |
| Post-PCI 48h ECG | |
| [postekg48:inline] | |
| Post-PCI 72h ECG | |
| [postekg72:inline] | |
| Does ECG show evolution compatible with acute myocardial infarction ? | <ul><li>Yes</li><li>No</li><li>Undefined</li></ul> |
| (Characteristic Q wave and/or ST normalization and/or T wave inversion) | ○ Undefined |
| . ( | |

## EKG modülü (ECG module) 2

| Study ID# | |
|---|---|
| You are viewing ECGs from the patient with the record number patient was admitted to [merkez] on [randomizasyon_tarihi]. | of [record_id], who is a [age] year-old [gender]. This |
| To access PMCardio App: https://difoccult.pmcardio.com | |
| The first pre-PCI ECG | |
| [ekg1:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | 3 |
| The second pre-PCI ECG | |
| [ekg2:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | ~(C) · (10) |
| The third pre-PCI ECG | |
| [ekg3:inline] | |
| Expert interpretation: | 4.65 |
| ○ OMI ○ not-OMI ○ Undefined | |
| The fourth pre-PCI ECG | |
| [ekg4:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | |
| The fifth pre-PCI ECG | |
| [ekg5:inline] | |
| Expert interpretation: | |
| ○ OMI ○ not-OMI ○ Undefined | |
| Are there any dynamic changes suggestive of OMI in pre-PCI ECGs ? | ○ Yes<br>○ No |
| (Dynamic ST-T changes, Q wave development) | ○ Undefined |
| The first post-PCI ECG | |
| [postpci_ekg:inline] | |



| Post-PCI 24h ECG | |
|---|---|
| [postekg24:inline] | |
| Post-PCI 48h ECG | |
| [postekg48:inline] | |
| Post-PCI 72h ECG | |
| [postekg72:inline] | |
| Does ECG show evolution compatible with acute myocardial infarction ? | <ul><li>Yes</li><li>No</li><li>Undefined</li></ul> |
| (Characteristic Q wave and/or ST normalization and/or T wave inversion) | ○ Undefined |
| . ( | |

# Anjiyografi (Angiography)

| Study ID# | |
|---|---|
| Did the patient undergo angiography ? | ○ Evet ○ Hayır |
| Date of angiogram (As day-month-year and hour:minute) | |
| Access site<br>(Vascular access site for primary PCI) | ○ Radial ○ Femoral |
| Angina relieved before angiography ? | ○ Yes ○ No ○ Unknown |
| ST-segment elevation on monitor relieved before angiography ? | ○ Yes ○ No ○ Unknown |
| Infarct-related artery | ○ None ○ LMCA ○ LAD ○ CX ○ RCA ○ Other or more than one |
| Enter the "other" artery (IM, intermediary artery; D, diagonal artery; OM, obtuse marginal artery etc.) | |
| Culprit looking lesion<br>(Select all that applies) | ☐ Total occlusion with an impression of being acute ☐ >90% diameter stenosis ☐ Presence of thrombus ☐ Contrast staining ☐ Irregular borders suggesting ulcerated plaque |
| TIMI flow level before PCI to culprit lesion | <ul> <li>TIMI 0, No perfusion</li> <li>TIMI 1, No perfusion but penetration (contrast penetrates past the lesion, but cannot reach distal coronary bed)</li> <li>TIMI 2, Partial perfusion (contrast reaches to distal vascular bed, but entry, filling and clearance are slower than other vessels)</li> <li>TIMI 3, Complete perfusion (distal flow and clearance are the same as those in other vessels)</li> </ul> |
| PCI to culprit lesion ? | ○ Evet ○ Hayır |
| TIMI flow level after PCI to culprit lesion | <ul> <li>TIMI 0, No perfusion</li> <li>TIMI 1, No perfusion but penetration (contrast penetrates past the lesion, but cannot reach distal coronary bed)</li> <li>TIMI 2, Partial perfusion (contrast reaches to distal vascular bed, but entry, filling and clearance are slower than other vessels)</li> <li>TIMI 3, Complete perfusion (distal flow and clearance are the same as those in other vessels)</li> </ul> |

| Additional lesions (Select for diameter stenosis of >30% for LMCA and 50% for other vessels. Do not include chronic total occlusion.) | ☐ LMCA ☐ LAD ☐ CX ☐ RCA ☐ Other lesions ☐ None |
|---|---|
| Enter other additional lesions<br>(IM, intermediary artery; D, diagonal artery; OM,<br>obtuse marginal artery etc. Multiple lesions should be<br>separated with commas) | |
| Vessels with chronic total occlusions (Do not include infarct-related artery.) | ☐ LMCA ☐ LAD ☐ CX ☐ RCA ☐ Other additional lesions |
| Enter other chronic total occlusions<br>(IM, intermediary artery; D, diagonal artery; OM,<br>obtuse marginal artery etc.) | 3 |
| Any additional PCI ? (The number vessels with non-culprit PCI at the same admission) | ○0 ○1 ○2 ○≥3 |

Since the patient is excluded, you do not need to fill this form.
(If you think this is an error, please check your answer for "Has the patient been excluded?" on the first form (Identification).)



# Hastanedeki klinik değişkenler (In-hospital clinical parameters)

| Study ID# |
|---|
| Upload post-PCI ECG<br>(if PCI not done, the first ECG at CCU) |
| Upload 24th hour ECG |
| Upload 48th hour ECG |
| Upload 72nd hour ECG |
| 24h troponin level (troponin level in ng/L [=pg/mL], e.g.; 12) |
| 48h troponin level (troponin level in ng/L [=pg/mL], e.g.; 12) |
| 72h troponin level (troponin level in ng/L [=pg/mL], e.g.; 12) |
| Ejection fraction (Percentage, e.g.; 55) |
| Wall motion score (Total point in 17-segment model, where 1=normokynesia, 2=hypokynesia, 3=akynesia) |
| Any other occlusion or re-occlusion during hospital Stay ? |

Since the patient is excluded, you do not need to fill this form. (If you think this is an error, please check your answer for "Has the patient been excluded?" on the first form (Identification).)



# Çıkış bilgileri (Clinical parameters on discharge)

| Study ID# | |
|---|---|
| Recommend allowing access for physicians to e-pulse account. (For easy access to long-term follow-up). | |
| In-hospital intubation after randomization | ○ Evet ○ Hayır |
| In-hospital cardiopulmonary resuscitation after randomization | ○ Evet ○ Hayır |
| In-hospital mortality after randomization | ○ Evet ○ Hayır |
| Final diagnosis (If preliminary diagnosis is confirmed, select "Myocardial infarction". If the patient was enrolled with a preliminary diagnosis of MI, but myocardial injury has been accounted for another reason later on, then select "Other troponin elevations". If no troponin rise observed, select "Other". If the patient died before any troponin result could be obtained, decide according to clinical scenario). | <ul> <li>Myocardial infarction</li> <li>Other troponin elevations (Heart failure, myocarditis, pulmonary embolism etc.)</li> <li>Other</li> </ul> |
| Aspirin<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
| P2Y12 inhibitors<br>(Prescribed medications on discharge) | <ul><li>○ None</li><li>○ Clopidogrel</li><li>○ Ticagrelor</li><li>○ Prasugrel</li></ul> |
| OAC/NOAC<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
| ACEI/ARB<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
| ARNI<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
| SGLT2i<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
| Beta-blocker<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
| Calcium channel blocker<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
| MRA (Prescribed medications on discharge) | ○ Evet ○ Hayır |



| Loop diuretic<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |
|--------------------------------------------------------|----------------|
| Statin<br>(Prescribed medications on discharge) | ○ Evet ○ Hayır |

Since the patient is excluded, you do not need to fill this form. (If you think this is an error, please check your answer for "Has the patient been excluded?" on the first form (Identification) or "In-hospital mortality?" in Discharge data form.)



#### Takip ve sonlanım (Long-term follow-up)

| Study ID# | |
|---|---|
| Long-term hospitalization<br>(Hospitalization in the first year) | ○ Evet ○ Hayır |
| Date of hospitalization<br>(The first hospitalization after discharge) | |
| Was the reason for hospitalization cardiovascular in origin ? | |
| Due to coronary by-pass surgery ?<br>(Direct transfer after index admission or planned<br>surgery after discharge) | ○ Evet ○ Hayır |
| Was the cause of admission PCI ? (Can be an elective or emergent admission.) | ○ Evet ○ Hayır |
| Was this PCI planned ?<br>(Can be an elective or emergent PCI.) | ○ Evet ○ Hayır |
| Long-term mortality<br>(Mortality in the first year after discharge) | ○ Evet ○ Hayır |
| Mortality date | |
| Was the reason for death cardiovascular in origin? | ○ Yes ○ No ○ Unknown |

You do not need to input any data to this form, since the patient has been excluded from the study. (If you think this message is inappropriate, check your response to "Has the patient been excluded?" (in Identification form).

